CLINICAL TRIAL: NCT05272202
Title: Study of Modulations of Motor Brain Activity Following Stimulation of the Median Nerve During General Anesthesia
Brief Title: Investigation of Cerebral Motor Activity Modulations Following Median Nerve Stimulation During General Anaesthesia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head of anesthesiology department, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STIM-MOTANA
Record Dates: First submitted 2022-01-11; First posted 2022-03-09 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Accidental Awareness During General Anesthesia
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Median nerve stimulation (Experimental)
  Interventions: Drug: Propofol; Device: Median nerve stimulation; Device: EEG measurements

INTERVENTIONS:
Drug: Propofol — STIM-MOTANA is an interventional and prospective study conducted in patients scheduled for surgery under general anesthesia, involving EEG measurements and median nerve stimulation. In this study, 30 patients will undergo surgery under total intravenous anesthesia using a propofol target-controlled infusion pump. The rest of the anesthetic protocol will be at the discretion of the anesthesiologist in charge. After surgery, patients will have a gradual decrease of propofol at different effect-site concentrations (from 4.0 μg/ml to 2.0 μg/ml, in increments of 0.5 μg/ml).
Device: Median nerve stimulation — The right-hand median nerve will be stimulated in the same way as for measurement with a conduction velocity or for an evoked potential. Two stimulation electrodes will be placed on the right-hand wrist according to the standards.The stimulation is transcutaneous and painless using the specific Micromed device Sd Ltm Stim Energy (Micromed, Mˆacon, France). The stimulus intensity will range between 3 and 14 mA. The stimulation duration will be 100 ms with a frequency of 0.1 Hz.
Device: EEG measurements — Changes in ERD and ERS patterns during median nerve stimulation according to the various propofol concentrations will be continuously monitored by an EEG amplifier. EEG signals will be acquired using the OpenViBE platform with a Biosemi Active Two 64-channel EEG system, arranged in the Biosemi's ABC system covering the entire scalp at 2048 Hz. Among all recorded sites, some of the electrodes will be localized around the primary motor cortex, the motor cortex, the somatosensory cortex, and the occipital cortex.

SUMMARY:
Accidental Awareness during General Anesthesia (AAGA) occurs in 1-2% of high-risk practice patients and is a cause of severe psychological trauma, termed post-traumatic stress disorder (PTSD). Actually, no monitoring techniques can accurately predict or detect an AAGA. Since the first reflex for a patient during an AAGA is to move, a brain-computer interface (BCI) based on the detection of an intention of movement would be conceivable to alert the anesthetist. The investigators previously showed that median nerve stimulation (MNS) could be the keystone of a BCI specialized in the detection of movement intention. Indeed, based on these previous results, the investigators can envisage a routine system where the patient would be stimulated at the median nerve position, while a BCI device would analyze the event-related desynchronization (ERD) and event-related synchronization (ERS) modulations in the motor cortex to check whether the patient is intending to move or not. According to the investigator's knowledge, no published studies have investigated the detection of EEG patterns in relation to peripheral nerve stimulation over the sensorimotor cortex during general anesthesia. The main objective of this study is to describe the changes in terms of ERD and ERS modulations, in the EEG signal over the motor cortex, during general anesthesia with propofol, while a median nerve stimulation is performed.

STIM-MOTANA is an interventional and prospective study conducted in patients scheduled for surgery under general anesthesia, involving EEG measurements and median nerve stimulation. In this study, 30 patients will undergo surgery under total intravenous anesthesia using a propofol target-controlled infusion pump. The rest of the anesthetic protocol will be at the discretion of the anesthesiologist in charge. Changes in ERD and ERS during median nerve stimulation according to the various propofol concentrations will be continuously monitored by an EEG amplifier. Pre- and post-injection comparisons of propofol will be performed by paired series tests. After surgery, patients will have a gradual decrease of propofol at different effect-site concentrations (from 4.0 μg/ml to 2.0 μg/ml, in increments of 0.5 μg/ml).

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years and <81 years
* Right-handed
* Programmed for surgery with the use of an intravenous anesthesia with a propofol concentration objective

Exclusion Criteria:

* Allergy to propofol, soy or peanuts
* BMI<20 or >30
* Pregnant or breastfeeding women
* Adult unable to give consent
* Medical or surgical history that may interfere with median nerve stimulation or the obtention of the EEG signal (for example: diabetes, polyneuropathy, central neurodegenerative disease, epilepsy, brain surgery)
* History of right median nerve injury
* Amputation of the upper right limb
* Impossibility of affixing an EEG helmet
* Addiction

Ages: 18 Years to 81 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Amplitude of the ERD (event-related desynchronization)/ERS (event- related synchronization) | From the time each stimulation is performed until 4 seconds after the stimulation is completed.
  The main evaluation outcome will be the amplitude of the ERD (event-related desynchronization)/ERS (event- related synchronization) after median nerve stimulation, within 4 s of the stimulation, at various propofol concentrations. This amplitude will be calculated using a baseline taken before each stimulation. The amplitudes of the ERD and ERS will be extracted. The ERDs and ERSs will be displayed from the time each stimulation is performed until 4 s after the stimulation is completed.

SECONDARY OUTCOMES:
Detection of ERD patterns via new machine-learning algorithms (percent of correct detection) | From the time each stimulation is performed until 4 seconds after the stimulation is completed.
  Verify the detection of ERD patterns via new machine-learning algorithms at different propofol concentrations. ERD patterns will be analysed manually, as well as automated by a machine-learning algorythm. Endpoint will be the percentage (%) of correctly identified ERD pattern by the algorythm.
Modulation of ERD patterns by anesthetics drugs. Percentage of variation in amplitude. | From the time each stimulation is performed until 4 seconds after the stimulation is completed.
  Another secondary criteria will to describe how the ERD generated by an MNS would be modulated by anesthetics drugs. Amplitude of ERD patterns will be recorded (microV) and the effect of anesthetic drugs on this amplitude will be described as percentage change.
Detection of ERS patterns via new machine-learning algorithms (percentage of correct detection) | From the time each stimulation is performed until 4 seconds after the stimulation is completed.
  Verify the detection of ERS patterns via new machine-learning algorithms at different propofol concentrations. ERS patterns will be analysed manually, as well as automated by a machine-learning algorythm. Endpoint will be the percentage (%) of correctly identified ERS pattern by the algorythm.
Modulation of ERS patterns by anesthetics drugs via new machine-learning algorithms (percentage change in amplitude) | From the time each stimulation is performed until 4 seconds after the stimulation is completed.
  Another secondary criteria will to describe how the ERS generated by an MNS would be modulated by anesthetics drugs. Amplitude of ERS patterns will be recorded (microV) and the effect of anesthetic drugs on this amplitude will be described as percentage change.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Schmartz, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rimbert S, Lelarge J, Guerci P, Bidgoli SJ, Meistelman C, Cheron G, Cebolla Alvarez AM, Schmartz D. Detection of Motor Cerebral Activity After Median Nerve Stimulation During General Anesthesia (STIM-MOTANA): Protocol for a Prospective Interventional Study. JMIR Res Protoc. 2023 Feb 2;12:e43870. doi: 10.2196/43870. PMID 36729587